CLINICAL TRIAL: NCT07395674
Title: Evaluation of the Effect of Subcutaneous Dexpanthenol Administration on Wound Epithelialization: A Pilot Randomized Controlled Study
Brief Title: Subcutaneous Dexpanthenol Administration and Wound Epithelialization
Acronym: DEXPAN-WOUND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dilara CANBAY OZDEMIR (Other)
Responsible Party: Sponsor-Investigator, Dilara CANBAY OZDEMIR, Assistant Professor of Family Medicine, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-FM-Dexpanthenol-2026
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Wounds; Diabetic Foot Ulcer; Venous Leg Ulcers; Arterial Ulcer
Keywords: Dexpanthenol; Chronic Wounds; Wound Healing; Epithelialization; Diabetic Foot Ulcer; Venous Leg Ulcer; Arterial Ulcer; Randomized Controlled Trial
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer | interventions — dexpanthenol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group and will remain in their assigned group throughout the study. Both groups will be followed in parallel according to the same visit schedule and assessment procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive standard wound care plus perilesional subcutaneous dexpanthenol injections administered at predefined intervals according to a standardized protocol.
  Interventions: Drug: Dexpanthenol; Other: Standard Wound Care
- Control Group (Active Comparator): Participants in this group will receive standardized wound care alone without subcutaneous dexpanthenol administration.
  Interventions: Other: Standard Wound Care

INTERVENTIONS:
Drug: Dexpanthenol — Dexpanthenol will be administered by perilesional subcutaneous injection around the wound area in addition to standard wound care. The injection dose and volume will be standardized according to wound size, with a limited number of treatment sessions.
  Arms: Intervention Group
Other: Standard Wound Care — Standard wound care includes wound cleansing with saline solution and topical wound management according to institutional protocols.

SUMMARY:
Chronic wounds are wounds that do not heal properly over time and can significantly reduce quality of life. Common types include diabetic foot ulcers, venous leg ulcers, and arterial ulcers. Improving wound healing and speeding up skin regeneration (epithelialization) are important goals in the care of these patients.

Dexpanthenol is a vitamin B5 derivative that supports skin repair and tissue regeneration. It is widely used in topical treatments, and injectable forms are approved for clinical use. However, the effects of subcutaneous (under the skin) dexpanthenol injections on chronic wound healing have not been sufficiently studied in clinical settings.

The purpose of this study is to evaluate whether adding subcutaneous dexpanthenol injections to standard wound care improves wound healing compared with standard wound care alone. Adult patients with non-infected chronic wounds will be randomly assigned to one of two groups. One group will receive standard wound care only, while the other group will receive standard wound care plus subcutaneous dexpanthenol injections around the wound area.

Wound healing will be assessed by measuring changes in wound size and the degree of skin epithelialization over time using standardized and objective methods. Safety will be monitored by recording local reactions at the injection site and any other adverse events during the study.

The results of this study may provide preliminary clinical evidence on the effectiveness and safety of subcutaneous dexpanthenol as an additional treatment option for chronic wound management.

DETAILED DESCRIPTION:
Chronic wounds, including diabetic foot ulcers, venous leg ulcers, and arterial ulcers, represent a major clinical challenge due to delayed healing, increased risk of complications, and reduced quality of life. Impaired epithelialization, prolonged inflammation, and insufficient tissue regeneration are key mechanisms contributing to non-healing wounds. Therefore, interventions that support epithelial repair and wound closure may improve clinical outcomes when added to standard wound care.

Dexpanthenol, a provitamin B5 derivative, is converted to pantothenic acid and plays an essential role in coenzyme A metabolism, which is involved in cellular energy production and tissue repair. Experimental and clinical studies have suggested that dexpanthenol may enhance fibroblast activity, epithelialization, and skin barrier restoration. Injectable formulations of dexpanthenol are approved for clinical use; however, data on subcutaneous administration for chronic wound healing are limited.

This study is designed as a randomized, open-label, controlled clinical trial to evaluate the effect of subcutaneous dexpanthenol administration on wound epithelialization when added to standard wound care. Adult patients with non-infected chronic wounds, including diabetic foot ulcers, venous leg ulcers, and arterial ulcers, will be enrolled. Eligible participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group using computer-generated block randomization.

Participants in the intervention group will receive standard wound care plus perilesional subcutaneous dexpanthenol injections administered at predefined intervals. The dose and injection volume will be standardized according to wound size, and a limited number of treatment sessions will be applied. Participants in the control group will receive standardized wound care alone. Both groups will follow the same visit schedule and assessment procedures throughout the study period.

Wound healing will be evaluated using objective and standardized methods. The primary outcome is the percentage change in wound area from baseline to follow-up visits. Secondary outcomes include changes in epithelialization percentage, time to complete epithelialization, wound bed tissue composition, and safety outcomes. Safety assessments will focus on local injection-site reactions and the occurrence of any adverse events, which will be systematically recorded during each visit.

This study aims to provide structured clinical data on the feasibility, safety, and potential clinical benefit of subcutaneous dexpanthenol as an adjunctive treatment in chronic wound management. The findings are expected to contribute to future studies and inform the design of larger-scale clinical trials in this field.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Presence of a chronic wound, including diabetic foot ulcer, venous leg ulcer, or arterial ulcer.
* Target wound size between 1 and 20 cm² at baseline.
* Non-infected wound, defined by the absence of purulent discharge, foul odor, spreading erythema, cellulitis, or systemic signs of infection.
* Clinically stable patients without the need for systemic antibiotic therapy.
* Ability to understand the study procedures and provide written informed consent.
* Willingness and ability to comply with study visits and treatment schedule.

Exclusion Criteria:

* Clinical signs of wound infection or requirement for systemic antibiotic treatment.
* Critical limb ischemia, defined as ankle-brachial index <0.5, rest pain, gangrene, or extensive tissue necrosis.
* Wounds exposing bone, tendon, or joint structures, or suspected osteomyelitis.
* Wound size smaller than 1 cm² or larger than 20 cm².
* Malignant, autoimmune, vasculitic, or specific dermatologic conditions causing the wound.
* Known hypersensitivity or allergy to dexpanthenol or any component of the study treatments.
* Pregnancy or breastfeeding.
* Cognitive impairment or inability to provide informed consent.
* Participation in another interventional clinical trial that could interfere with the outcomes of this study.
* Any medical condition that, in the investigator's judgment, could compromise participant safety or study integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Wound Area | Baseline (Day 0) to Day 19 ±1 and Day 26 ±1
  The primary outcome measure is the percentage change in wound area from baseline. Wound area will be calculated using standardized ruler-based measurements of the longest length and widest width of the wound and applying an elliptical area formula. The percentage change in wound area will be calculated by comparing baseline measurements with follow-up measurements.

SECONDARY OUTCOMES:
Change in Wound Epithelialization Percentage | Baseline (Day 0) to Day 19 ±1 and Day 26 ±1
  Wound epithelialization will be assessed as the percentage of epithelial tissue covering the wound surface. Changes in epithelialization percentage over time will be evaluated using standardized wound bed tissue composition assessments.
Time to Complete Epithelialization | Up to approximately 26 days
  Time to complete epithelialization will be defined as the number of days from baseline to the first visit at which the wound shows complete epithelial coverage without drainage, confirmed at two consecutive follow-up visits.
Wound Bed Tissue Composition | Baseline (Day 0) to Day 26 ±1
  Wound bed tissue composition, including percentages of epithelial tissue, granulation tissue, and fibrin or necrotic tissue, will be assessed at each study visit using standardized clinical evaluation methods.
Local Injection Site Reactions and Adverse Events | Baseline (Day 0) to Day 26 ±1
  Safety outcomes will include the assessment of local injection site reactions such as pain, erythema, edema, induration, and nodule formation, as well as the occurrence of any other adverse events recorded throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Canbay Özdemir, MD, Principal Investigator — Ordu University Faculty of Medicine, Department of Family Medicine
Locations (1):
- Ordu University Training and Research Hospital, Ordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Heise R, Skazik C, Marquardt Y, Czaja K, Sebastian K, Kurschat P, Gan L, Denecke B, Ekanayake-Bohlig S, Wilhelm KP, Merk HF, Baron JM. Dexpanthenol modulates gene expression in skin wound healing in vivo. Skin Pharmacol Physiol. 2012;25(5):241-8. doi: 10.1159/000341144. Epub 2012 Jun 29. PMID 22759998
- [Background] Proksch E, de Bony R, Trapp S, Boudon S. Topical use of dexpanthenol: a 70th anniversary article. J Dermatolog Treat. 2017 Dec;28(8):766-773. doi: 10.1080/09546634.2017.1325310. Epub 2017 May 14. PMID 28503966
- [Background] Gorski J, Proksch E, Baron JM, Schmid D, Zhang L. Dexpanthenol in Wound Healing after Medical and Cosmetic Interventions (Postprocedure Wound Healing). Pharmaceuticals (Basel). 2020 Jun 29;13(7):138. doi: 10.3390/ph13070138. PMID 32610604
- [Background] Metin N, Karapinar T, Turan C. Lip mesotherapy with dexpanthenol in the treatment of isotretinoin-induced cheilitis. J Cosmet Dermatol. 2022 Oct;21(10):4684-4690. doi: 10.1111/jocd.14993. Epub 2022 May 10. PMID 35426210